CLINICAL TRIAL: NCT03288311
Title: Protocolized Post-Extubation Respiratory Support (PROPER) Study
Brief Title: Protocolized Post-Extubation Respiratory Support Study
Acronym: PROPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Casey, Pulmonary and Critical Care Medicine Research Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 170650
Record Dates: First submitted 2017-09-15; First posted 2017-09-20 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Mechanical Ventilation Complication; Acute Respiratory Failure; Intubation Complication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocolized Post-extubation Respiratory Support (Active Comparator): Qualifying patients undergoing extubation in an ICU bed randomized to post-extubation respiratory support will receive either non-invasive ventilation or high flow nasal cannula (as determined by a prespecified protocol and applied by a respiratory therapist) from the time of extubation until 5AM the following morning
  Interventions: Other: Protocolized post-extubation respiratory support
- Usual Care (Active Comparator): Qualifying patients undergoing extubation in an ICU bed randomized to usual care will receive standard-of-care treatment, which may include post-extubation respiratory support at the discretion of their clinical team.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Protocolized post-extubation respiratory support — Qualifying patients undergoing extubation in an ICU bed randomized to post-extubation respiratory support will receive either non-invasive ventilation or high flow nasal cannula (as determined by a prespecified protocol and applied by a respiratory therapist) from the time of extubation until 5AM the following morning
  Arms: Protocolized Post-extubation Respiratory Support
Other: Usual Care — Qualifying patients undergoing extubation in an ICU bed randomized to usual care will receive standard-of-care treatment, which may include post-extubation respiratory support at the discretion of their clinical team.
  Arms: Usual Care

SUMMARY:
Invasive mechanical ventilation is common in the medical intensive care unit, and the period of time following extubation remains high risk as 11 to 15% of patients require reintubation after their first extubation. Reintubation is associated with increased rates of nosocomial infection and is an independent predictor of mortality. Non-invasive ventilation and high flow nasal cannula are the only therapies that have been shown to reduce the rate of reintubation. Recent clinical trials suggest that all patients might benefit from some form of post-extubation respiratory support, but use of these therapies in usual care remains low. PROPER is a cluster-randomized, multiple-crossover trial comparing a respiratory therapist driven protocol to provide post-extubation respiratory support to all patients, compared to usual care. The trial will enroll patients undergoing extubation in the Medical ICU at Vanderbilt from October 2017 until March 2019. The primary outcome will be reintubation within 96 hours.

DETAILED DESCRIPTION:
PROPER is a prospective, pragmatic, cluster-randomized, multiple-crossover trial comparing a respiratory therapist driven protocol for post-extubation respiratory support to usual care. The primary outcome will be reintubation by 96 hours. All adults (age 18 or older) who receive at least 12 hours of mechanical ventilation and are extubated in the Vanderbilt Medical ICU will be enrolled in the trial. The ICU will be divided into 2 clusters, based on the geographic areas covered by the two respiratory therapist dedicated to that ICU. The study will occur in three month blocks. One cluster will be randomized to receive protocolized post-extubation respiratory support (as prescribed by a protocol and delivered by a respiratory therapist), while the other cluster receives usual care, which can include post-extubation respiratory support when requested by the clinical team. At the end of three months, the clusters will cross-over, such that each cluster will spend half of the study receiving protocolized post-extubation respiratory and half of the study receiving usual care. It is anticipated that approximately 630 patients will be enrolled from the medical ICU during the 18 month study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is located in a participating unit
2. Patient undergoing extubation from mechanical ventilation
3. Patient has been receiving mechanical ventilation for at least 12 hours
4. Age ≥ 18 years old

Exclusion Criteria:

1. Patient is receiving ventilation via a tracheostomy
2. Patient is being extubated to comfort measures or has "Do Not Reintubate" order in place at the time of extubation
3. Patient has required reintubation after a prior attempt at extubation during this hospitalization
4. Unplanned or self-extubation, where immediate reintubation is deemed necessary by the clinical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd W Rice, MD, MSc, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available following publication of the primary trial results
Access Criteria: Data dictionary will be available upon requests. Requests for deidentified patient-level data will be reviewed by the trial steering committee. Sharing of deidentified data will require approval of proposed secondary analysis and a signed data use agreement.

REFERENCES:
- [Derived] Casey JD, Vaughan EM, Lloyd BD, Billas PA, Jackson KE, Hall EJ, Toporek AH, Buell KG, Brown RM, Richardson RK, Rooks JC, Buie RB, Wang L, Lindsell CJ, Ely EW, Self WH, Bernard GR, Rice TW, Semler MW. Protocolized Postextubation Respiratory Support to Prevent Reintubation: A Randomized Clinical Trial. Am J Respir Crit Care Med. 2021 Aug 1;204(3):294-302. doi: 10.1164/rccm.202009-3561OC. PMID 33794131
- [Derived] Casey JD, Vaughan ER, Lloyd BD, Bilas PA, Hall EJ, Toporek AH, Buell KG, Brown RM, Richardson RK, Rooks JC, Wang L, Lindsell CJ, Ely EW, Self WH, Bernard GR, Rice TW, Semler MW; Pragmatic Critical Care Research Group. Protocolized Post-Extubation Respiratory Support to prevent reintubation: protocol and statistical analysis plan for a clinical trial. BMJ Open. 2019 Aug 2;9(8):e030476. doi: 10.1136/bmjopen-2019-030476. PMID 31377713

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
Started | 359 | 392
Completed | 359 | 392
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care | Total
Number analyzed (Participants) | 359 | 392 | 751
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [43 to 66] | 57 [42 to 66] | 57 [42 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 187 | 342
  Male | 204 | 205 | 409
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 287 | 317 | 604
  Black or African American | 58 | 59 | 117
  Asian | 3 | 8 | 11
  Other | 5 | 4 | 9
  Not Reported | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Reintubation
Description: Any placement of an endotracheal tube for any indication within 96 hours of extubation, censored at the first of hospital discharge or 96 hours after extubation
Time Frame: within 96 hours of extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
Number analyzed (Participants) | 359 | 392
Participants | 57 | 52

2. Secondary Outcome: All-cause In-hospital Death
Description: All cause mortality, censored at the first of hospital discharge or 28 days after extubation
Time Frame: from extubation to discharge or 28 days post-extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
Number analyzed (Participants) | 359 | 392
Participants | 29 | 41

3. Secondary Outcome: ICU-free Days
Description: number of days alive from final ICU transfer until study day 28
Time Frame: from extubation to discharge or 28 days post-extubation
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
Number analyzed (Participants) | 359 | 392
days | 26 [23 to 26] | 26 [22 to 26]

4. Secondary Outcome: Ventilator-free Days
Description: number of days alive from final invasive mechanical ventilation until study day 28
Time Frame: from extubation to discharge or 28 days post-extubation
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
Number analyzed (Participants) | 359 | 392
days | 28 [28 to 28] | 28 [28 to 28]

5. Secondary Outcome: Time to Reintubation
Description: Time from extubation to reintubation
Time Frame: from extubation to discharge or 28 days post-extubation
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
Number analyzed (Participants) | 359 | 392
hours | 56 [21 to 147] | 47 [18 to 163]

6. Secondary Outcome: Number of Patients Requiring Re-intubation for Respiratory Indication
Description: Number of patients in each group with respiratory indication for reintubation.
Time Frame: within 96 hours of extubation
Population: Full trial population
Measure: Count of Participants; unit: Participants
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
Number analyzed (Participants) | 359 | 392
Participants | 35 | 33

7. Secondary Outcome: Number of Patients Requiring Reintubation for Laryngeal Edema
Description: Percentage of patients in each group with laryngeal edema as the indication for reintubation
Time Frame: within 96 hours of extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
Number analyzed (Participants) | 359 | 392
Participants | 0 | 2

8. Secondary Outcome: Number of Patients With Delirium
Description: As defined by Confusion Assessment Method for the ICU (CAM-ICU) score and reported by bedside nurse. A report of "Yes" indicates the presence of delirium, which is reflected in the reported cases.
Time Frame: within 96 hours of extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
Number analyzed (Participants) | 359 | 392
Participants | 160 | 151

9. Secondary Outcome: Number of Patients With Agitation
Description: As defined by RAS score and reported by bedside nurse
Time Frame: within 96 hours of extubation
Population: Data was unavailable for collection
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Lowest S/F Ratio
Description: Lowest ratio of O2 saturation to concentration inhaled oxygen (FIO2)
Time Frame: between 0-6 hours, 6-12 hours, and 12-24 hours after extubation
Measure: Median (Inter-Quartile Range); unit: ratio of O2 saturation to concentration
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
Number analyzed (Participants) | 359 | 392
ratio of O2 saturation to concentration
  0-6 hours | 237.5 [205.0 to 254.3] | 268.5 [224.4 to 344.4]
  6-12 hours | 242.5 [222.5 to 303.3] | 318.5 [240.0 to 438.1]
  12-24 hours | 242.5 [214.6 to 340.7] | 327.6 [240.0 to 438.1]

11. Secondary Outcome: Highest Respiratory Rate
Description: Highest respiratory rate
Time Frame: between 0-6 hours, 6-12 hours, and 12-24 hours after extubation
Measure: Median (Inter-Quartile Range); unit: breaths per minute
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
Number analyzed (Participants) | 359 | 392
breaths per minute
  0-6 hours | 23 [20 to 28] | 24 [21 to 28]
  6-12 hours | 24 [19 to 28] | 24 [20 to 29]
  12-24 hours | 25 [21 to 30] | 25 [21 to 29]

12. Secondary Outcome: Use of High Flow Nasal Cannula (HFNC) or Non-invasive Ventilation (NIV) Beyond 24 Hours Post-extubation
Description: Use of non-invasive ventilation or high flow nasal cannula beyond 24 hours post-extubation
Time Frame: from 24 hours post extubation to 96 hours post-extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
Number analyzed (Participants) | 359 | 392
Participants | 26 | 14

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to 28 days after enrollment
Description: Because this trial compared strategies commonly used in routine clinical care, the only events that were recorded or reported as adverse events were those that were related to the study and serious or unexpected. Patients who require mechanical ventilation in the critical care setting are at risk for hypoxemia, hypotension, cardiac arrest, and death. These events were recorded as study outcomes and only recorded as AEs if related to the study intervention, which was expected to be rare.
Arm/Group | Protocolized Post-extubation Respiratory Support | Usual Care
All-Cause Mortality (participants affected / at risk) | 29/359 | 41/392
Serious Adverse Events (participants affected / at risk) | 0/359 | 0/392
Other Adverse Events (participants affected / at risk) | 0/359 | 0/392

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT03288311/Prot_SAP_000.pdf